CLINICAL TRIAL: NCT05411133
Title: A Phase 1, First-in-human Study of Cabotamig (ARB202), Bispecific Antibody to CDH17 and CD3 in Advanced Gastrointestinal Malignancies
Brief Title: Treatment of Cabotamig (ARB202) in Advanced Gastrointestinal Cancer Patients
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Arbele Pty Ltd (Industry)
Responsible Party: Sponsor
Organization: Arbele Limited (Industry)
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: A001
Record Dates: First submitted 2022-05-25; First posted 2022-06-09 (Actual); Last update posted 2025-09-04 (Actual); Status verified 2025-08

CONDITIONS: Gastrointestinal Cancer; Cholangiocarcinoma; Liver Cancer; Colorectal Adenocarcinoma; Pancreatic Cancer; Gastric Cancer; Esophageal Adenocarcinoma; Gastroesophageal Junction; Gastrointestinal Neuroendocrine Tumors
MeSH Terms: conditions — Gastrointestinal Neoplasms; Cholangiocarcinoma; Liver Neoplasms; Pancreatic Neoplasms; Stomach Neoplasms; Adenocarcinoma Of Esophagus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (5):
- Phase 1a: Dose Escalation (Experimental)
  Interventions: Drug: Cabotamig (ARB202)
- Phase 1b: Low dose Cabotamig (ARB202) (Experimental)
  Interventions: Drug: Cabotamig (ARB202)
- Phase 1b: High dose Cabotamig (ARB202) (Experimental)
  Interventions: Drug: Cabotamig (ARB202)
- Phase 1b: Low dose Cabotamig (ARB202) + Immune Checkpoint Inhibitor (Experimental)
  Interventions: Drug: Cabotamig (ARB202)
- Phase 1b: High dose Cabotamig (ARB202) + Immune Checkpoint Inhibitor (Experimental)
  Interventions: Drug: Cabotamig (ARB202)

INTERVENTIONS:
Drug: Cabotamig (ARB202) — Cabotamig (ARB202), Atezolizumab

SUMMARY:
This study aims to find out:

1. The tolerability of Cabotamig (ARB202) in adults with advanced solid gastrointestinal tumors who failed the standard treatment. People can participate if their tumor has the CDH17 marker.
2. To find out how study drug is broken down in the body
3. To know the effects of the study drug on the tumor.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed colorectal, pancreatic, gastric adenocarcinoma, primary liver cancer or metastatic liver disease, or cholangiocarcinoma that is metastatic or unresectable and for which standard curative or palliative measures do not exist or are no longer effective.
* Malignancies should possess with ≥10% expression of CDH17 confirmed by immunohistochemistry except for CRC patients. If the testing is based on fine-needle aspiration (FNA) biopsy, the patient will be considered eligible when tumor aspirate demonstrates detectable positive staining cells for CDH17.
* Eastern Cooperative Oncology Group (ECOG) performance status of ≤2.
* Life expectancy > 3 months.
* Measurable disease as defined by RECIST 1.1 criteria
* Blood coagulation parameters:

  * PT INR ≤ 1.5X ULN
  * PTT INR ≤1.2X ULN
* Patients must have adequate venous peripheral access for apheresis.
* Satisfactory organ and bone marrow function as defined by:

  * absolute neutrophil count > 1,000/μL
  * platelets >100,000/μL
  * hemoglobin ≥9 g/dL
  * serum ALT and AST ≤ 3X ULN or AST and ALT ≤5X ULN, if liver function abnormalities are thought to be from underlying malignancy
  * total serum bilirubin ≤ 2X ULN
  * Creatinine <1.5X ULN
  * Stable amylase for 2 weeks

Exclusion Criteria:

* Prior gene therapy or therapy with any murine monoclonal antibodies or any murine containing product.
* Concurrent treatment with any anticancer agent including chemotherapy, hormonal therapy or radiation therapy. Must be 5 X half-life or 6 weeks (whichever is shorter) post dosing of previous cancer therapies.
* History of allergy or hypersensitivity to murine proteins or study product excipients
* Females who are pregnant, trying to become pregnant, or breastfeeding.
* Diagnosis of HIV or chronic active viral hepatitis (HBV, HCV, HIV).
* Active infection requiring systemic treatment.
* Active brain, leptomeningeal, or paraspinal metastases, except for asymptomatic metastases and are stable on a steroid dose of ≤ 10mg/day of prednisone or its equivalent for at least 14 days prior to the start of study interventions.
* Impaired cardiac function (AHA NY Heart Association Grade II-IV) or clinically significant cardiac disease.
* Lack of recovery of prior CTCAE Grade 3 or above adverse events due to earlier therapies.
* Chronic use of corticosteroids in excess of >10mg daily of prednisone or equivalent within 4 weeks prior to alopecia.
* Concomitant use of complementary or alternative medication or therapy such as Chinese herbal medicine.
* History of Crohn's disease, inflammatory bowel disease, or ulcerative colitis within the past 5 years
* Abnormal bowel function which would make assessment of bowel permeability difficult to access
* Major trauma or major surgery within 4 weeks prior to first dose of study drug

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Estimated)
Dates: Start 2022-05-30 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Incidence and severity of adverse events | 8 weeks post initial dose

SECONDARY OUTCOMES:
Amount of Cabotamig (ARB202) in plasma after single and multiple doses of ARB202 (Cabotamig) in patients | 16 weeks
Biochemical and physiological effects of Cabotamig (ARB202) on the amount of circulating ARB202 (Cabotamig) level in patients | 16 weeks
Biochemical and physiological effects of Cabotamig (ARB202) on the amount of soluble CDH17 level in patients | 16 weeks
Biochemical and physiological effects of Cabotamig (ARB202) on the amount IL-2 level in patients | 16 weeks
Effect of Cabotamig (ARB202) on tumour as determined by changes in RECIST evaluation from baseline | 6 weeks

CONTACTS AND LOCATIONS:
Locations (3):
- Australia (2):
  - Southern Oncology Clinical Research Unit, Adelaide
  - St George Private Hospital, Sydney
- Queen Mary Hospital, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No